CLINICAL TRIAL: NCT02545413
Title: Randomized,Double-blind, Placebo Controlled Trial to Study the Efficacy and Safety of Probiotics in Adult Patients With Irritable Bowel Syndrome-diarrhea Predominant (IBS-D)
Brief Title: Study to Determine Efficacy of Probiotics in Irritable Bowel Syndrome
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Investigator (Dr Amit) not interested to carry out the study
Sponsor: Next Gen Pharma India Pvt. Ltd. (Industry)
Collaborators: Department of Gastroenterology, Govt. Medical College, Kozhikode, Kerala, India (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRC/2015/protocol/24
Record Dates: First submitted 2015-08-31; First posted 2015-09-10 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-03

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic (Experimental): Probiotic VSL#3 will be given at a dose of one capsule thrice daily for 8 weeks, amounting to a total of 337.5 billion CFU/day. Each capsule contains 112.5 billion viable lyophilized bacteria of four strains of Lactobacillus (L. acidophilus DSM 24735, L. plantarum DSM 24730, L. paracasei DSM 24733, L. delbrueckii subsp. bulgaricus DSM 24734), three strains of Bifidobacterium (B. longum DSM 24736, B. breve DSM 24732, B. infantis DSM 24737) and one strain of Streptococcus (S. thermophilus DSM 24731) and excipients.
  Interventions: Drug: Probiotic VSL#3
- Placebo (Placebo Comparator): Placebo capsules will be given at a dose of one capsule thrice daily for 8 weeks; Placebo capsules contain all excipients as present in capsules (without the 8 strains of bacteria as mentioned above).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Probiotic VSL#3
  Arms: Probiotic
Drug: Placebo
  Arms: Placebo

SUMMARY:
Irritable bowel syndrome (IBS) is the most common functional GI disorder in which abdominal pain and/or discomfort is associated with changes in bowel habit, and with features of disordered defecation. IBS affects 10-20% of the population and causes a marked reduction of quality of life in affected individuals.The high prevalence of IBS is accompanied by large societal economic burdens and negative effects on the quality of life in affected patients. It is divided into 3 types IBS-D diarrhea predominant, IBS-C constipation predominant, IBS-M mixed sub type.

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS) is the most common functional GI disorder affecting 10-20% of the population and causing a marked reduction of quality of life in affected individuals. An altered brain-gut axis has been accepted as a main pathogenetic mechanism of IBS, which is associated with a dysfunction of the GI autonomic nervous system. These alterations may lead to abnormal visceral hypersensitivity and aberrations of gut motility. Recently, additional potential mechanisms of IBS have emerged including alteration of gut microbiota and low-grade inflammation/immune activation. These factors might lead to abnormal motility and visceral hypersensitivity and contribute to the symptoms. Naïve gut microbiota plays important roles in the maintenance of gut homeostasis by direct bactericidal effects and the evolution of both innate and adaptive immune systems. Gut microbiota is thought to play important roles in the pathogenesis of IBS. This is evident from the fact that IBS occurs more frequently after intestinal infection or antibiotics treatment. Studies have shown that the alterations of the intestinal microbiota are observed in IBS patients.Considering the relationship between alteration of gut microbiota and inflammation of gut, manipulation of gut microbiota by probiotics appears to be an ideal treatment modality for IBS. However, the beneficial effects and efficacy of altering gut microbiota by probiotics to improve the symptoms of IBS have not been consistent in clinical trials and therefore it remains uncertain as an effective treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Positive diagnoses of IBS subtype IBS-D defined by Rome III criteria, and who meet the following criteria:

   a) Abdominal Pain Intensity: weekly average of worst daily (in past 24 hours) b) abdominal pain score of > 3.0 on a 0 to 10 point scale & c) Stool Consistency of at least one stool with a consistency of Type 6 or Type 7 Bristol stool score (BSS) on at least 2 days per week
2. Signed informed consent

Exclusion Criteria:

1. Patients currently using non-steroidal anti-inflammatory drugs, corticosteroids and mast cell stabilizers, or topical or systemic antibiotics in the past 1 month.
2. Patients with major abdominal surgery, a history of inflammatory bowel disease or diverticular disease, celiac disease (by detection of anti-transglutaminase and anti-endomysial antibodies), allergic diseases, including asthma (excluded by family and personal history and specific anti-IgE antibodies), and other organic or psychiatric disorders as assessed by medical history, appropriate consultations and laboratory tests.
3. Females who are Pregnant, breast-feeding, or not using reliable methods of contraception

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-05; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of the intensity of abdominal pain relief and change in stool consistency before and after treatment, between the two arms | 8 wks (after end of treatment)
  The defecation component of the primary endpoint will be evaluated by assessing stool consistency as per "Bristol Stool Form Scale". Abdominal pain component of primary end point will be accessed by using an 11-point (i.e., 0 to 10) numeric rating scale that asks patients daily to rate their worst abdominal pain over the past 24-hours

SECONDARY OUTCOMES:
Comparison of Quality of Life parameters as measured by IBS-QoL Questionnaire before and after treatment, between the 2 arms | 8 wks (after end of treatment) and 20 weeks (12 weeks after end of follow-up period; at end of study)
Comparison of Quality of Life parameters as measured by SF-36 Questionnaire before and after treatment, between the 2 arms | 8 wks (after end of treatment) and 20 weeks (12 weeks after end of follow-up period; at end of study)
Comparison of Visceral hypersensitivity/Rectal sensitivity before and after treatment between the two arms | 8 wks (after end of treatment)
  Visceral hypersensitivity/Rectal sensitivity as measured between and within arms using a lubricated rectal balloon catheter for the duration taken for first defecation, first instance of pain and the pain threshold

CONTACTS AND LOCATIONS:
Overall Officials: Shejal A Hanmant, DM Trainee, Principal Investigator — Government Medical College, Kozhikide, Kerala, India; Varghese Thomas, DM, Principal Investigator — Government Medical College, Kozhikide, Kerala, India
Locations (1):
- Department of Gastroeneterology, Government Medical College, Kozhikode, Kerala, India